CLINICAL TRIAL: NCT05983406
Title: Role of Doppler Endoscopic Probe in the Diagnosis of Subepithelial Gastrointestinal Lesions.
Acronym: DopplerSEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Francisco Baldaque-Silva (Other)
Responsible Party: Sponsor-Investigator, Francisco Baldaque-Silva, MD PhD, Senior consultant, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KarolinskaUH 2019-05404; 2019-05404 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Subepithelial Tumors of the Upper Gastrointestinal Tract
Keywords: Doppler, EUS, SEL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Doppler endoscopic probe in the diagnosis of subepithelial gastrointestinal lesions
  Interventions: Device: Doppler investigation

INTERVENTIONS:
Device: Doppler investigation — Doppler investigation

SUMMARY:
RESEARCH PLAN I-TITLE Role of Doppler endoscopic probe in the diagnosis of subepithelial gastrointestinal lesions.

II-BACKGROUND Subepithelial lesions (SEL) are commonly encountered during routine endoscopies with an estimated prevalence of 3.5%. Most of the SELs are detected during upper gastrointestinal endoscopy. Subsequently, endoscopic ultrasound (EUS) is performed to better characterize the lesion and to rule out the presence of a vascular lesion before tissue sampling due to the high risk of severe bleeding with tissue acquisition in vascular injury. However, EUS can rarely establish a definitive diagnosis per se with limited accuracy.

In large lesions, it is possible to use cytology or histology needles via the EUS instrument to collect cells/tissue within the lesion. It can lead to accurate diagnosis and consistent management. However, EUS-guided tissue sampling can be technically challenging, with poor yield for small or mobile SELs. In addition, EUS is an expensive technique, high operator dependency and performed only in tertiary centers. It creates a time gap between endoscopic detection and the EUS examination and increases costs. That delay in diagnosis is a source of anxiety for the patient and for the caregivers.

Several methods were proposed to increase the diagnostic yield of tissue acquisition techniques, such as "bite-on-bite" biopsies which showed a limited diagnostic yield. Alternatively, the "unroofing" technique has also been advocated for histological diagnosis. In unroofing, a loop is used to remove the normal epithelium covering the subepithelial lesions and after epithelial removal, a biopsy forceps or loop is used to sample subepithelial lesions. Other techniques include endoscopic resection by snare or submucosal dissection. These enable a surgical specimen but are technically demanding and have been complicated by perforation and bleeding in most series.

There is a need for a method that enables rapid diagnosis in the same session as endoscopic detection of SEL regardless of their size. That method should ideally enable histological diagnosis with low risks of complications and should not require high technical expertise and should not be highly dependent on the operator. The ideal solution to address the diagnosis of gastrointestinal (GI) SEL would be one that would provide a tissue sampling after exclusion of a highly vascular lesion, in the same session as endoscopic detection.

Doppler endoscopic probe (DEP) is a Doppler endoscopic probe specially developed for the GI system, which enables blood flow detection during endoscopy.

DEP is CE and FDA approved and can be used through the working channel of the endoscope. Unlike standard EUS, which requires advanced endoscopic training, DEP is much easier to use. It allows the characterization of lesions as non-vascular, venous or arterial. Recent studies have demonstrated the safety and efficacy of DEP in vascular characterization in the gastrointestinal tract.

III PURPOSE

Primary objective:

* Proof of concept evaluation of the role of DEP in the characterization of GI SEL as non-vascular or vascular (arterial or venous)
* Relationship between findings on DEP versus findings on EUS (considered the gold standard) regarding SEL characterization as non-vascular or vascular (arterial or venous).

Secondary purposes:

* Accuracy in removing the histological characterization of subepithelial GI lesions.
* Complications in connection with tissue acquisition
* Inter-observer agreement of DEP and EUS results. IV METHODS This is a pilot projective feasibility study that will be run by Karolinska University Hospital in Stockholm Patients with subepithelial GI lesions were referred for EUS evaluation. The study will include 30 patients.

A conventional gastroscopy will be performed. After identification of the lesion, DEP is performed. The DEP probe is lubricated and deployed through the working channel of the endoscope. The probe will contact the mucosa slightly, covering the SEL. Then evaluate the lesion in 2 different angels. The results will be characterized and recorded qualitatively: no flow / arterial flow / venous flow and in terms of intensity: soft, medium or high.

After DEP, evaluation EUS will be performed by another endoscopist who will be tied to the DEP results. EUS will be considered the gold standard.

After both assessments, the lesion is characterized as no vessel / arterial / venous and as soft / medium / high flow intensity.

EUS will be followed by removal of SEL in patients where EUS excludes the presence of high vessel disease. "Unroofing" will be performed using a conventional endoscopic loop, through the working channel of the endoscope. After the surface of the lesion is disturbed, a biopsy forceps will be used for tissue acquisition. Tissue will be stored in formalin and processed and evaluated by the pathologist.

DETAILED DESCRIPTION:
RESEARCH PLAN

I-TITLE Role of doppler endoscopic probe in the diagnosis of subepithelial gastrointestinal lesions.

II-BACKGROUND

Subepithelial lesions (SELs) are commonly encountered on routine endoscopies with estimated prevalence of 3.5% (PMID: 24238309). Most small SELs are asymptomatic and benign, but their pathological diagnosis may be challenging, and sometimes impossible with conventional technology.

Most of SELs are detected during upper gastrointestinal endoscopy. Afterwards, endoscopic ultrasound (EUS) is usually performed in order to better characterize the lesion and to exclude the presence of a vascular lesion. EUS enables evaluation of the size, structure and location of the lesion within the GI wall (submucosa/muscularis mucosa/ submucosa/muscularis propria), but can seldom stablish a definitive diagnosis per se. EUS provides valuable information regarding the layer of origin and can suggest a diagnosis, but it has been shown to have limited accuracy. (PMID: 12190103).

In lesions larger than 2cm, it is possible to use dedicated cytologi (FNA) or histology (FNB) needles thought the EUS instrument in order to collect cells/tissue from within the lesion. That may lead to proper diagnosis and consequent management. However, EUS-guided tissue sampling can be technically challenging, with poor yields for small or mobile SELs (20306384). Additionally, EUS is an expensive technique, highly operator dependent and usually only performed in tertiary centers. That creates a time gap between the endoscopic detection and the EUS investigation, and increases the costs. That delay in the diagnosis is a source of anxiety for the patient and for health care providers alike.

In cases with small or mobile SEL, in which a definitive diagnosis cannot be stablished with EUS plus FNA/FNB, surveillance is recommended. But the later, is associated with high costs and high burden for the health care system.

Several methods were advocated to increase the diagnostic yield of tissue acquisition techniques such as "bite- on-bite" forceps biopsy that showed a limited diagnostic yield (PMID: 12518134), with one prospective study showing a diagnostic yield of only 17% compared with 87% with endoscopic resection (PMID: 16813799). Alternatively, unroofing technique has also been advocated in this context. With unroofing a snare is used to remove the normal epithelium that is covering the subepithelial lesion, and after epithelial removal a biopsy forceps is used to sample the subepithelial lesion. Other techniques include endoscopic resection by snaring or submucosal dissection. These enable a surgical specimen but are technically demanding and have been complicated by perforation and bleeding in most series.

Although endoscopic resection may have the advantage of providing both a complete pathological diagnosis as well as treatment for the tumor in selected patients, it is questionable whether endoscopic resection of the entire lesion is needed for diagnostic purposes, because of the associated long procedure time and potentially serious complications, such as bleeding and perforation.

EUS is usually performed before biopsy sampling, snaring or endoscopic resection in order to exclude the presence of a highly vascular SEL, due to the high risk of severe bleeding in case of tissue acquisition in a vascular lesion.

There is a need for a method that would enable rapid diagnosis in the same session as endoscopic detection of SELs irrespective of their size. That method should ideally enable histological diagnosis with low risks of complications and should not demand high technical expertise and should not be highly operator dependent. The ideal solution to address the diagnosis of gastrointestinal (GI) SEL would be one that would provide a tissue sampling after exclusion of a highly vascular lesion, in the same session as the endoscopic diagnosis.

Doppler endoscopic probe (DEP) is a 2-mm diameter, single-use, Doppler endoscopic probe (Vascular Technology Inc, Nashua, NH) specifically developed for GI tract, that enables blood flow detection during endoscopy. As lesions are unlikely to bleed substantially without a major supply of blood flow, the applicability of endoscopic DEP resides in the ability to detect blood flow within submucosal blood vessels that feed a potentially bleeding lesion within the GI tract.

DEP is CE and FDA approved and may be used through the working channel of the endoscope. The DEP system is a 20-MHz, pulsed-wave Doppler ultrasound unit with 3 preset scanning depths: from the surface to 1.5, 4, and 7 mm. It has an audible Doppler output signal but does not have a visual monitor display. The unit is portable and battery-powered. Unlike standard EUS, which requires advanced endoscopic training, DEP is much more straightforward to use (15557966). The applicability of endoscopic Doppler US resides in the ability to detect blood flow within submucosal blood vessels that feed a potentially bleeding lesion within the GI tract. A positive DEP signal has been defined as a repetitive and similar visual spiking waveform (or audible signal) of at least 3 consecutive cycle duration (indicating pulsatile blood flow and minimizing the chance of a false-positive signal) (PMID: 10968843).

Recent studies had demonstrated the safety and efficacy of DEP in the vascular characterization of gastrointestinal peptic ulcers (26318834, 28167214).

III- AIMS

Primary aims:

* Proof-of-concept evaluation of the role of DEP in the characterization of GI SEL as highly vascular or non-highly vascular.
* Correlation between findings on DEP versus finding on EUS (considered the gold standard) in terms of SEL characterization as highly vascular or non-highly vascular.

Secondary aims:

* Accuracy of unroofing in the histological characterization of subepitelial GI lesions.
* Complications associated with tissue acquisition through unroofing technique such as bleeding or perforation
* Inter-observer agreement of the DEP findings.

IV- METHODS

STUDY DESIGN

This is a pilot prospective feasibility study that will be run by Karolinska University Hospital in Stockholm

STUDY POPULATION Patients with subepithelial GI lesions referred for EUS evaluation. The study will include 20 patients.

Inclusion criteria

- Presence of subepithelial lesion on the GI tract.

Exclusion criteria

* Anticoagulation therapy that cannot be discontinued
* Liver cirrhosis with coagulopathy or varices
* Malignancy

All patients will receive a detailed explanation regarding the procedure, its risks, benefits, and alternatives, and provided written informed consent before inclusion (Appendix 1).

Participants clinical, demographic, and procedural information will be obtained and recorded at enrollment (Appendix 2).

Patients under antiplatelet or anticoagulant drugs will be handled according to published guidelines.

OUTCOME PARAMETERS PRIMARY OUTCOME PARAMETERS DEP. The auditory sound from arterial flow corresponds to a sound like a blood pressure "swish-swish," whereas venous flow is a low-pitched venous hum. Intensity will be recorded as soft, medium, or loud.

Doppler on EUS will be evaluated as standard using the color-doppler and also wave flow assessment.

SECONDARY OUTCOME PARAMETERS Adverse events are defined as any complication in which DEP, EUS, unroofing or related procedures are a contributing factor and include bleeding and perforation.

Perforation is defined as a full thickness breach in the GI wall with or without symptoms.

Intraprocedural bleeding is considered significant and a complication when:

* blood transfusion is needed
* premature termination of endoscopic occurs

Delayed bleeding is defined as clinical evidence of bleeding manifested by melena or hematochezia from up to 14 days after the procedure that demanded presentation to the emergency department, hospital admission or medical intervention.

Adverse events are classified as:

* acute (during procedure)
* early (<48 h)
* late (>48 h).

In terms of severity they are characterized as:

* mild (unplanned medical assistance, hospital admission, hospitalization <3 days, hemoglobin drop <3 g, no transfusion)
* moderate (4-10 days hospitalization, <4 units blood transfusion, repeat endoscopic intervention, radiological intervention)
* severe (hospitalization >10 days, intensive care unit (ICU) admission, need for surgery, >4 units blood transfusion) or fatal (death attributable to procedure) [7, 8].

ENDOSCOPIC PROTOCOL

A conventional gastroscopy will be performed. After identification of the lesion, DEP will be performed. The DEP probe will be lubricated and deployed through the working channel of the endoscope. The probe will contact slightly the mucosa covering the SEL. Then will evaluate the lesion in 2 different angels (one at the top and one at the base of the lesion). First, the superficial Doppler depth setting (< 1.5 mm) will be used, followed by the middle setting (< 4 mm). Assessment will be recorded and endoscopist diagnosis (arterial flow/venous flow, soft/medium/loud intensity) will be registered. All DEP will be performed by the same endoscopist (MO). Findings will be characterized and registered qualitatively: no flow/arterial flow/venous flow and in terms of intensity: soft, medium, or loud.

After DEP, evaluation EUS will be performed by another endoscopists (FBS) that will be blinded to the DEP findings. EUS will be considered the gold standard.

After both assessments the lesion will be characterized as no vascular/low vascular/highly vascular flow.

EUS will be followed by unroofing of the SEL in patients in which EUS excluded the presence of a highly vascular lesion. Unroofing will be performed using a conventional endoscopic snare, through the working channel of the endoscope. After the surface of the lesion is unroofed, a biopsy forceps will be used for tissue acquisition. Tissue will be stored in formalin and processed and evaluated by pathologist.

All data will be registered. All procedures will be recorded in video and audio (DEP).

POST PROCEDURE PROTOCOL

Before Discharge After unroofing, patients will be closely monitored for 2-4 hours under continuous monitoring and then discharged if no complications detected.

After Discharge At week 8 after discharge, patients will have a hospital visit for assessment of complications and control endoscopy.

V-SIGNIFICANCE With this study it will be possible to evaluate the strategy of DEP and unroofing in the assessment of GI SEL. In case of positive results: good accuracy in the diagnosis/exclusion of vascular lesions with DEP and good histological yield with unroofing, this strategy may be further validated and might change the paradigm of management of GI SEL.

ELIGIBILITY:
Inclusion Criteria:

* Presence of subepithelial lesion on the GI tract.

Exclusion Criteria:

* Anticoagulation therapy that cannot be discontinued
* Liver cirrhosis with coagulopathy or varices
* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
DEP accuracy | From enrollment to the end of study at 8 weeks
  DEP. The auditory sound from arterial flow corresponds to a sound like a blood pressure "swish-swish," whereas venous flow is a low-pitched venous hum. Intensity will be recorded as soft, medium, or loud. Doppler on EUS will be evaluated as standard using the color-doppler and also wave flow assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital & Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunt GC, Smith PP, Faigel DO. Yield of tissue sampling for submucosal lesions evaluated by EUS. Gastrointest Endosc. 2003 Jan;57(1):68-72. doi: 10.1067/mge.2003.34. PMID 12518134
- [Background] Philipper M, Hollerbach S, Gabbert HE, Heikaus S, Bocking A, Pomjanski N, Neuhaus H, Frieling T, Schumacher B. Prospective comparison of endoscopic ultrasound-guided fine-needle aspiration and surgical histology in upper gastrointestinal submucosal tumors. Endoscopy. 2010 Apr;42(4):300-5. doi: 10.1055/s-0029-1244006. Epub 2010 Mar 19. PMID 20306384
- [Background] Rosch T, Kapfer B, Will U, Baronius W, Strobel M, Lorenz R, Ulm K; German EUS Club. Endoscopic ultrasonography. Accuracy of endoscopic ultrasonography in upper gastrointestinal submucosal lesions: a prospective multicenter study. Scand J Gastroenterol. 2002 Jul;37(7):856-62. PMID 12190103
- [Background] Binmoeller KF, Shah JN, Bhat YM, Kane SD. Suck-ligate-unroof-biopsy by using a detachable 20-mm loop for the diagnosis and therapy of small subepithelial tumors (with video). Gastrointest Endosc. 2014 May;79(5):750-5. doi: 10.1016/j.gie.2013.09.028. Epub 2013 Nov 12. PMID 24238309